CLINICAL TRIAL: NCT00084071
Title: Tifacogin (Recombinant Tissue Factor Pathway Inhibitor) for the Treatment of Patients With Severe Community-Acquired Pneumonia
Brief Title: Tifacogin for the Treatment of Patients With Severe Community-Acquired Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTFP561A2308
Record Dates: First submitted 2004-06-04; First posted 2004-06-08 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2012-07

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Tifacogin

INTERVENTIONS:
Drug: Tifacogin

SUMMARY:
The purpose of this study is to determine whether tifacogin is effective and safe in the treatment of patients with severe community-acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of community-acquired pneumonia supported by additional clinical, radiological, and microbiological evidence
* Pneumonia of sufficient severity to require ICU admission and management

Exclusion Criteria:

* Pregnancy
* Weight over 150 kg
* Patients at increased risk of bleeding
* Treatment with drotrecogin alfa or anticipated need for drotrecogin alfa
* Treatment with heparin or anticipated need for heparin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2136 (Actual)
Dates: Start 2004-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Compare the effect of tifacogin vs placebo administration.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (150):
- United States (51):
  - Mobile, Alabama
  - Loma Linda, California
  - Los Angeles, California
  - Orange, California
  - Sacramento, California
  - San Diego, California
  - San Jose, California
  - Denver, Colorado
  - Farmington, Connecticut
  - New Haven, Connecticut
  - Newark, Delaware
  - Bay Pines, Florida
  - Clearwater, Florida
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - Atlanta, Georgia
  - Conyers, Georgia
  - Decatur, Georgia
  - Chicago, Illinois
  - Oak Park, Illinois
  - Muncie, Indiana
  - New Albany, Indiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Cumberland, Maryland
  - Detroit, Michigan
  - Southfield, Michigan
  - St Louis, Missouri
  - Butte, Montana
  - Reno, Nevada
  - Buffalo, New York
  - Johnson City, New York
  - Greensboro, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Allentown, Pennsylvania
  - Pawtucket, Rhode Island
  - Providence, Rhode Island
  - Spartanburg, South Carolina
  - Knoxville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Winchester, Virginia
  - Seattle, Washington
  - Tacoma, Washington
- Argentina (4):
  - Mar del Plata, Buenos Aires
  - Tandil, Buenos Aires
  - Tres de Febrero, Buenos Aires
  - Capital Federal
- Australia (15):
  - Garran, Australian Capital Territory
  - Camperdown, New South Wales
  - Kingswood, New South Wales
  - Cairns, Queensland
  - Nambour, Queensland
  - Southport, Queensland
  - Woodville, South Australia
  - Hobart, Tasmania
  - Launceston, Tasmania
  - Box Hill, Victoria
  - Footscray, Victoria
  - Heidelburg, Victoria
  - Parkville, Victoria
  - Nedlands, Western Australia
  - Perth, Western Australia
- Belgium (10):
  - Brussels, Jette
  - Bouge
  - Braine-l'Alleud
  - Brussels
  - Ghent
  - Liège
  - Mons
  - Ottignies
  - Seraing
  - Yvoir
- Brazil (10):
  - Fortaleza, Ceará
  - Belgium, Salvador, Estado de Bahia
  - Salvador, Estado de Bahia
  - Curitiba, Paraná
  - Recife, Pernambuco
  - Pelotas, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Florianópolis, Santa Catarina
  - Campinas, São Paulo
  - São José do Rio Preto, São Paulo
- Canada (13):
  - Calgary, Alberta
  - Edmonton, Alberta
  - New Westminster, British Columbia
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - Kingston, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Montreal, Quebec
- Chile (2):
  - Santiago
  - Temuco
- France (9):
  - Argenteuil
  - Belfort
  - Besançon
  - La Roche Sur Yoon
  - Limoges
  - Paris
  - Pierre-Bénite
  - Saint-Michel
  - Tours
- Germany (3):
  - Lübeck
  - München
  - Regensburg
- Malaysia (5):
  - George Town
  - Johor Bahru
  - Kota Bharu Kelantan
  - Kuala Lumpar
  - Kuala Selangor
- Netherlands (3):
  - 's-Hertogenbosch
  - Rotterdam
  - Utrecht
- New Zealand (4):
  - Grafton, Auckland
  - Otahuhu, Auckland
  - Christchurch
  - Hastings
- Lima, Peru
- Singapore, Singapore
- South Africa (6):
  - KwaKhangela, Durban
  - Parktown, Johannesburg
  - Bloemfontein
  - Centurion
  - Kimberley
  - Parktown West
- South Korea (6):
  - Wŏnju, Gangwon-do
  - Namdong-gu, Incheon
  - Gyeonggi-do
  - Gyunggi
  - Seoul
  - Suwon
- Spain (4):
  - Sabadell, Barcelona
  - Madrid
  - Palma de Mallorca
  - Santiago de Compostela
- United Kingdom (3):
  - Glasgow
  - Livingston
  - London

REFERENCES:
- [Derived] Laterre PF, Opal SM, Abraham E, LaRosa SP, Creasey AA, Xie F, Poole L, Wunderink RG. A clinical evaluation committee assessment of recombinant human tissue factor pathway inhibitor (tifacogin) in patients with severe community-acquired pneumonia. Crit Care. 2009;13(2):R36. doi: 10.1186/cc7747. Epub 2009 Mar 15. PMID 19284881
- See also: Results for CTFP561A2308 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3160